CLINICAL TRIAL: NCT04102085
Title: the Study of Persistent Organic Pollutants in Human Milk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tse Lap Ah, Associate professor, Chinese University of Hong Kong
Other Study IDs: DH/SEB/NCD/18/2018-19
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Breast Milk Collection
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Breast milk
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mothers under 30: no intervention will be administered
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The study aims to recruit eligible participants and conduct interviews, collect human milk samples, and conduct laboratory analysis of persistent organic pollutants' levels in human milk samples.

DETAILED DESCRIPTION:
Persistent Organic Pollutants (POPs) are a group of chemicals which have been intentionally or inadvertently produced and introduced into the environment. Due to their stability and transport properties, they are widely distributed around the world, and are even found in places where they had never been used, such as the arctic regions. Given their long half-lives and fat solubility, POPs tend to bioaccumulate in animals, particularly in long-lived species at the top of the food-chain. POPs appear at higher concentrations in fat-containing foods, including fish, meat, eggs and milk. POPs are also present in the human body and traces can be found in human milk. The most commonly mentioned POPs are organochlorine pesticides, such as DDT, industrial chemicals, most notably polychlorinated biphenyls (PCBs), and by-products, especially polychlorinated dibenzodioxins (PCDDs) and polychlorinated dibenzofurans (PCDFs). As a group, POPs are of concern for both the environment and human health 1.

With the ratification of the Stockholm Convention on POPs in early 2004, the international community signaled its commitment to reduce or eliminate production and emission of POPs into the environment and ultimately, the human body. There were 12 POPs initially listed under the Convention in 2004 2. The Convention is effective to the People's Republic of China, including the Hong Kong Special Administrative Region (HKSAR). The Environmental Protection Department (EPD) coordinates the HKSAR Government's efforts for the Convention and prepared the HKSAR Implementation Plan 3, in which the Department of Health (DH) is required to conduct the regular local monitoring of POPs in human milk.

The first study of POPs in human milk by DH was conducted during 2008 to 2011, which was made reference to Guidelines for Developing a National Protocol of the Fourth World Health Organization (WHO) - Coordinated Survey of Human Milk for POPs in Cooperation with United Nations Environment Programme (UN Environment) (2007) 4.

Results of the first study by DH was published in a scientific journal 5 and submitted to EPD, which were also discussed in the HKSAR Implementation Plan for the Stockholm Convention on POPs (2016) 5. Compared to the related earlier local studies 7,8,9 conducted by local universities, levels of POPs in human milk had declined over time.

Mothers should be reassured that breast milk is naturally the superior food for infants. The study is intended to provide data to evaluate the effectiveness of the international agreement, i.e. the Stockholm Convention, which aims to reduce the levels of certain POPs in our environment.

The study will also support national capabilities for monitoring and sound management of POPs.

ELIGIBILITY:
Inclusion Criteria:

* Primiparae;
* 30 years of age or below;
* Have normal pregnancy;
* Breastfeeding one infant only, and not multiple pregnancy;
* Resided in Hong Kong for at least 10 years immediately before the date of interview;
* Available for sample collection within 3 to 8 weeks of delivery; and
* Both mother and child should be apparently healthy and free from any known infectious or other diseases (e.g. clinical hepatitis, AIDs, HIV).

Exclusion Criteria:

* participants with previously diagnosed major diseases such as hepatitis, AIDS and other such diseases shall be excluded from the study

Max Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Primiparae
Study Population: Fifty eligible participants (nursing mothers) will be identified during their postnatal visits at four selected Maternal Child Health Centres (MCHCs) of the Department of Health, representing four major regions in Hong Kong:
  Sai Ying Pun MCHC (Hong Kong Island); Kowloon City MCHC (Kowloon); Madam Yung Fung Shee MCHC (New Territories West); and Ma On Shan MCHC (New Territories East).
  If the recruitment is unsatisfactory in the above four centres, other MCHCs will be involved.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-09-25 (Estimated); Study Completion 2021-10-25 (Estimated)

PRIMARY OUTCOMES:
Amount of persistent organic pollutants in breast milk | 2 years
  Approximately 30 types of persistent organic pollutants will be tested

CONTACTS AND LOCATIONS:
Overall Officials: Lap Ah Tse, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Bonnie Kwok, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No